CLINICAL TRIAL: NCT04479592
Title: Colonoscopy is an Aerosol-generating Procedure and Water-immersion Technique May Decrease the Amount of Aerosol Generated
Brief Title: Colonoscopy is an Aerosol Generating Procedure
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, CHAN SHANNON MELISSA, Assistant Professor, Chinese University of Hong Kong
Other Study IDs: 2020.200.2
Record Dates: First submitted 2020-07-17; First posted 2020-07-21 (Actual); Last update posted 2020-07-21 (Actual); Status verified 2020-07

CONDITIONS: To See if Colonoscopy is an Aerosol-generating Procedure and to Identify Ways to Minimise the Aerosol Generated
Keywords: Colonoscopy; Aerosol-generating procedure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Particle counter — Particle counter to measure the aerosol generated

SUMMARY:
With a commercially available particle counter, we can differentiate the particle counts of different sizes in different areas of the endoscopy room. An increase from baseline particles of < 5um during or after the procedure would suggest that the procedure is an AGP.

In this study, the particle counter from Met One Instruments model GT-526S will be used. A particle sizer is placed within 10cm of the anus, at the level of the endoscopists' face and at the level of the endoscopy nurse assistant's face The change in the particles of different sizes would be simultaneously recorded. The results of these three locations are compared to baseline and compared with each other

DETAILED DESCRIPTION:
Currently, the term droplet is often taken to refer to droplets >5 microns (μm) in diameter that fall rapidly to the ground under gravity, and therefore are transmitted only over a limited distance (e.g. ≤1 m). In contrast, the term droplet nuclei refers to droplets ≤5 μm in diameter that can remain suspended in air for significant periods of time, allowing them to be transmitted over distances >1 metre. With a commercially available particle counter, we can differentiate the particle counts of different sizes in different areas of the endoscopy room. An increase from baseline particles of < 5um during or after the procedure would suggest that the procedure is an AGP.

In this study, the particle counter from Met One Instruments model GT-526S will be used. The study will be conducted in the Prince of Wales Hospital endoscopy centre. A particle sizer is placed within 10cm of the anus, at the level of the endoscopists' face and at the level of the endoscopy nurse assistant's face The change in the particles of different sizes would be simultaneously recorded. The results of these three locations are compared to baseline and compared with each other.

ELIGIBILITY:
Inclusion Criteria:

- All patients who are planned for colonoscopy in the Prince of Wales Hospital, Hong kong

Exclusion Criteria:

* Patients where a flexible sigmoidoscopy was plannned Patients where the procedure was done in a negative pressure room Patients where the procedure was done in an endoscopy room other than the designated rooms Patients where the procedure was done under general anaesthesia

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients who are planned for colonoscopy in the Prince of Wales Hospital, Hong kong.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2020-06-01 (Actual); Primary Completion 2020-12-30 (Estimated); Study Completion 2021-01-31 (Estimated)

PRIMARY OUTCOMES:
Concentration of aerosol generated during the procedure | During the procedure
  Concentration of aerosol generated during the procedure

CONTACTS AND LOCATIONS:
Overall Officials: Shannon M Chan, FRCSEd, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Prince of Wales Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No